CLINICAL TRIAL: NCT01195142
Title: Adipose Tissue Gene Expression Profiles in Women With PCOS Versus Controls Matched for BMI
Brief Title: Adipose Tissue Gene Expression Profiles in Women With Polycystic Ovary Syndrome (PCOS) Versus Controls
Status: Completed | Type: Observational
Sponsor: The Adelaide and Meath Hospital (Other)
Collaborators: University College Dublin (Other)
Responsible Party: Dr James Gibney, AMNCH
Other Study IDs: DDC-UCD-ATCS
Record Dates: First submitted 2010-09-02; First posted 2010-09-06 (Estimated); Last update posted 2010-09-06 (Estimated); Status verified 2008-07

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PCOS-CSAT: Women with PCOS
- Control-CSAT: Control population consisting of women without PCOS, matched for age and BMI with the PCOS cohort

SUMMARY:
Adipose tissue is a central organ in mediating metabolic health. There is some evidence that women with polycystic ovary syndrome (PCOS) have a degree of adipose tissue dysfunction which may negatively affect their metabolic health. The aim of this study was to assess transcriptomic profiles of subcutaneous adipose tissue of women with PCOS in comparison with a control population matched on the basis of age and body mass index (BMI). A secondary aim was to then relate these gene expression profiles to the biochemical environment.

DETAILED DESCRIPTION:
Adipose tissue is a central organ in mediating metabolic health. There is some evidence that women with polycystic ovary syndrome (PCOS) have a degree of adipose tissue dysfunction which may negatively affect their metabolic health. The aim of this study was to assess transcriptomic profiles of subcutaneous adipose tissue of women with PCOS in comparison with a control population matched on the basis of age and body mass index (BMI). A secondary aim was to then relate these gene expression profiles to the biochemical environment.

ELIGIBILITY:
Inclusion Criteria:

* Had a positive diagnosis of PCOS as defined according to the NIH criteria as chronic oligomenorrhoea (< 9 menstrual cycles per year) and clinical and/or biochemical evidence of hyperandrogenism, in the absence of other disorders causing the same phenotype. Clinical criteria included hirsutism with a Ferriman-Galwey score greater than 9, acne or male pattern alopecia; biochemical criteria included total-testosterone, androstenedione or dehydroepiandrosterone sulphate (DHEAS) greater than the laboratory reference range.
* Were between the ages of 18 and 40

Exclusion Criteria:

* Were under 18 years or greater than 40 years old,
* Were non-Caucasian
* Were pregnant, lactating or trying to conceive
* Had a body mass index (BMI) <18kg/m2 or >50kg/m2
* Had a recent illness or any chronic illness likely to influence results
* Were taking hormonal contraception

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women with PCOS and a control population of women matched for age and body mass index (BMI)
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2007-12; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Transcriptomic profiling of subcutaneous adipose tissue of women with PCOS and age and BMI matched controls | Recruitment ran from Dec 2007-July 2008. Subjects attended the study location fasting on one occasion
  Gene expression profiles from women with PCOS and controls matched for age and BMI were determined by microarray analysis of whole subcutaneous adipose tissue samples. Single gene changes as well as pathway analyses will be used to determine differently expressed genes and pathways between the PCOS cohort and controls.

SECONDARY OUTCOMES:
Measurement of biomarkers of metabolic health (lipid, inflammatory markers) in plasma of PCOS cases and controls | Recruitment ran from Dec 2007-July 2008. Subjects attended the study location fasting on one occasion
  Biomarkers of metabolic health were assessed in plasma of women with PCOS and age and BMI matched controls. Lipid profile, hormonal profile, various key inflammatory markers and adipokines will be measured. Glucose and insulin concentrations will be assessed also. All parameters will be assessed following a 12 hour over night fast at the study location.

CONTACTS AND LOCATIONS:
Overall Officials: James Gibney, Dr, Principal Investigator — The Adelaide and Meath Hospital; Helen M Roche, Dr, Principal Investigator — University College Dublin
Locations (2):
- Ireland (2):
  - Diabetes Day Centre, The Adelaide and Meath Hosptial, Dublin, Dublin
  - Nutrigenomics Group, University College Dublin, Dublin, Leinster